CLINICAL TRIAL: NCT00926731
Title: A Phase I, Open-label, Multi-centre, Multiple Ascending Dose Study to Assess the Safety and Tolerability of AZD1152 in Combination With Low Dose Cytosine Arabinoside (LDAC) in Patients With Acute Myeloid Leukaemia (AML)
Brief Title: Study to Assess the Safety and Tolerability of AZD1152 in Combination With Low Dose Cytosine Arabinoside (LDAC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Paul K. Stockman, MBChB, PhD, Medical Science Director (Emerging Products Team II), AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1531C00018
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukaemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 2-((3-((4-((5-(2-((3-fluorophenyl)amino)-2-oxoethyl)-1H-pyrazol-3-yl)amino)quinazolin-7-yl)oxy)propyl)(ethyl)amino)ethyl dihydrogen phosphate; Cytarabine

ARMS (1):
- 1 (Experimental): AZD1152 variable dose in combination with 20 mg of LDAC. (The LDAC is given twice daily.)
  Interventions: Drug: AZD1152; Drug: LDAC (low dose cytosine arabinoside)

INTERVENTIONS:
Drug: AZD1152 — Variable dose via a 7-day continuous infusion
Drug: LDAC (low dose cytosine arabinoside) — 20 mg subcutaneous injection given twice daily

SUMMARY:
A study to assess the safety and tolerability of AZD1152 in combination with low dose cytosine arabinoside (LDAC) in patients with acute myeloid leukaemia (AML). The first three patients to complete a 28 day cycle in the cohort, before the second three patients start treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patient.
* Provision of written informed consent.
* De Novo (primary) or Secondary AML.
* Not eligible for intensive induction chemotherapy because of medical, social or psychological reasons.

Exclusion Criteria:

* Patients with AML of FAB M3 classification Acute Promyelocytic Leukaemia (APL).
* Patients with blast crisis of chronic myeloid leukaemia.
* Persistent, chronic, clinically significant toxicities from any prior anti- cancer therapy greater than CTCAE Grade 1 (except alopecia).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety as measured by Adverse Events, Vital Signs, ECGs, Clinical Chemistry, Haematology and Urinalysis | Information on these will be collected from the time of informed consent is signed, throughout the study.

SECONDARY OUTCOMES:
Assessment of the pharmacokinetics of AZD1152, its active moiety AZD1152 hQPA, and LDAC. | During the first treatment cycle for AZD1152, pre-dose and Days 2, 3,7, 8, 9, 10, 15 and 22. For LDAC, Days 7 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, Study Director — AstraZeneca; Hagop Kantarjian, Principal Investigator — M. D. Anderson, (University of Texas)
Locations (4):
- United States (2):
  - Research Site, Cleveland, Ohio
  - Research Site, Houston, Texas
- France (2):
  - Research Site, Le Chesnay
  - Research Site, Villejuif

REFERENCES:
- [Derived] Kantarjian HM, Sekeres MA, Ribrag V, Rousselot P, Garcia-Manero G, Jabbour EJ, Owen K, Stockman PK, Oliver SD. Phase I study assessing the safety and tolerability of barasertib (AZD1152) with low-dose cytosine arabinoside in elderly patients with AML. Clin Lymphoma Myeloma Leuk. 2013 Oct;13(5):559-67. doi: 10.1016/j.clml.2013.03.019. Epub 2013 Jun 10. PMID 23763917
- [Derived] Quintas-Cardama A, Ravandi F, Liu-Dumlao T, Brandt M, Faderl S, Pierce S, Borthakur G, Garcia-Manero G, Cortes J, Kantarjian H. Epigenetic therapy is associated with similar survival compared with intensive chemotherapy in older patients with newly diagnosed acute myeloid leukemia. Blood. 2012 Dec 6;120(24):4840-5. doi: 10.1182/blood-2012-06-436055. Epub 2012 Oct 15. PMID 23071272